CLINICAL TRIAL: NCT03238066
Title: A Prospective Phase II Study of Salvage Brachytherapy in Combination With Interstitial Hyperthermia for Locally Recurrent Prostate Carcinoma Following External Beam Radiation Therapy
Brief Title: Salvage Brachytherapy and Interstitial Hyperthermia for Locally Recurrent Prostate Carcinoma Following Radiation Therapy
Acronym: Prostata-BT-HT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Vratislav Strnad, Assistant Medical Director of the Dept. of Radiooncology, University of Erlangen-Nürnberg Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prostata-BT-HT
Record Dates: First submitted 2015-12-01; First posted 2017-08-03 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): The physician can choose either HDR or PDR brachytherapy.
  If HDR BT is chosen:
  d1: hyperthermia (IHT) 60 minutes + 10Gy HDR brachytherapy (HDRBT) d22: IHT 60 minutes + 10 Gy HDRBT d43: IHT 60 minutes + 10 Gy HDRBT
  If PDR BT is chosen:
  d1-3: IHT 60 minutes + 30Gy PDRBT d29-31: IHT 60 minutes + 30Gy PDRBT
  Interventions: Radiation: Brachytherapy; Other: Hyperthermia

INTERVENTIONS:
Radiation: Brachytherapy — HDR/PDR brachytherapy
Other: Hyperthermia — Interstitial hyperthermia

SUMMARY:
Salvage brachytherapy in combination with interstitial hyperthermia for locally recurrent prostate carcinoma following external beam radiation therapy.

DETAILED DESCRIPTION:
Salvage brachytherapy in combination with interstitial hyperthermia for locally recurrent prostate carcinoma following external beam radiation therapy:

Salvage brachytherapy: HDRBT: 3 x 10 Gy specified on prostate capsule/tumor margin (d1, 22, 43) or PDRBT: 2 x 30 Gy specified on prostate capsule/tumor margin (d1-3, 29-31) Hyperthermia: prostate heated to 40 - 47˚C for 30-60 minutes (60 minutes recommended) prior to brachytherapy dose delivery. Maximum temperature in surrounding critical normal organs should not exceed 43˚C

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed locally recurrent prostate cancer - biopsy performed < 6 months before registration;
* Histology: Adenocarcinoma, every Gleason score (2-10)
* Initial treatment (EBRT) completed > 24 months prior to biopsy;
* Androgen deprivation therapy for prostate cancer should be discontinued at least 3 months prior to patient registration
* Staging performed within 12 weeks prior to registration:

  * Local stage evaluated by DRE, TRUS or - if necessary - mpMRI (T1b, T1c, T2a, T2b, T2c, T3a, T3b);
  * Negative lymph nodes by imaging studies (at least one of these: choline PET scan, pelvic ± abdominal CT or MRI) or by lymphadenectomy (cN0 or pN0);
  * Negative bone scan (M0);
* PSA-DT > 6 months (PSA measurements taken of the 12 months prior to registration)
* Zubrod Performance Scale 0-2 (Appendix V) International Prostate Symptoms Score (IPSS) < 20 (Appendix VI), the IPSS score can be evaluated in patient on alpha-blockers;
* Baseline gastrointestinal (GI) or genitourinary (GU) toxicity grade 0-1 as defined in Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

In TRUS volume study performed 0-4 weeks before registration patient meets eligibility criteria for prostate brachytherapy as follows:

* Prostate/tumor volume <60ml
* The distance rear prostate edge - rectal mucosa >5mm
* Interference of pubic arch ruled out
* If local stage T3b: it must be possible to cover by the brachytherapy dose cancer infiltration

  * Prostate lenght (from apex plane to base plane) ≤ 45mm (technical criterion for 915 MHz frequency antennas)
  * The patient is suitable for spinal or general anesthesia
  * Age > 18 y.
  * Life expectancy > 5 years
  * absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
  * The patient must sign a study-specific informed consent form before study registration

Exclusion Criteria:

* Severe, active comorbidities:

  * Decompensated congestive heart disease
  * Chronic obstructive pulmonary disease exacerbation, respiratory failure
  * Hepatic insufficiency resulting in coagulation defects or clinical jaundice
* Other active malignancy or treatment of invasive or hematological malignancy
* Evidence of extraprostatic disease at local recurrence:

  * Local stage T4
  * Histologic or radiologic evidence of lymph node metastases (N1 or pN1)
  * Presence of distant metastases (M1)
* Any of the following prior therapies:

  * TURP within 6 months prior to registration
  * Prostatic salvage cryosurgery performed at least 6 months before registration
  * HIFU performed at least 6 months before registration
  * Androgen deprivation therapy within 3 months prior to registration
* Baseline gastrointestinal (GI) or genitourinary (GU) toxicity grade ≥ 2 as defined in Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Rate of late GI/GU grade 3 and more toxicities | up to 60 Months in Follow up

SECONDARY OUTCOMES:
Rate of acute GI/GU treatment-related adverse events | up to 24 months after start of recruitment
Time to biochemical failure | up to 60 Months in Follow up
  defined rise of PSA
Overall survival | up to 60 Months in Follow up
Disease-free survival | up to 60 Months in Follow up
Disease-specific survival | up to 60 Months in Follow up
Clinical patterns of tumor recurrence | up to 60 Months in Follow up

CONTACTS AND LOCATIONS:
Overall Officials: Vratislav Strnad, MD, Principal Investigator — Assistant Medical Director of the Dept. of Radiooncology
Locations (3):
- Strahlenklinik im Universitaetsklinikum Erlangen, Erlangen, Germany
- Poland (2):
  - Centrum Radiotherapii, Krakow
  - Maria Sklodowska-Curie Institute - Oncology Center, Warsaw